CLINICAL TRIAL: NCT02218658
Title: The Bioequivalence Between WE 941 OD Tablets (0.25mg as the Basis) Taken Without Water and Brotizolam Conventional Tablets (Lendormin® Tablets, 0.25 mg as the Basis) Taken With Water, as a Single Administration in Healthy Adult Male Subjects (Open-labelled, 2-way Cross-over Study)
Brief Title: Bioequivalence Between WE 941 OD and Brotizolam (Lendormin®) in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 263.507
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — brotizolam

ARMS (2):
- WE 941 OD (Experimental)
  Interventions: Drug: WE941 OD tablets
- Brotizolam (Active Comparator)
  Interventions: Drug: Brotizolam

INTERVENTIONS:
Drug: WE941 OD tablets
  Arms: WE 941 OD
Drug: Brotizolam
  Other Names: Lendormin®
  Arms: Brotizolam

SUMMARY:
The bioequivalence of WE 941 OD tablets prepared in oral disintegrating tablet form taken without water and brotizolam conventional tablets (Lendormin® tablets) taken with water, was evaluated in healthy adult male subjects (open-labelled, 2-way cross-over study)

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years
* Weight between 50 and 80 kg
* Obesity level within the range of +/- 20% of the standard weight according to the Body Mass Index (BMI) method
* Judged as eligible as a study object following the screening test by the investigator
* Volunteers to participate in the study, who are capable of giving written informed consent

Exclusion Criteria:

* Known hypersensitivity to drugs
* History of drug or alcohol abuse
* Received other investigational drug within 4 months of the trial drug administration
* Had > 400 mL of whole blood drawn within 3 months of the trial drug administration
* Had > 400 mL of blood components drawn within 1 month of the trial drug administration
* Used any drug within 10 days of the trial drug administration
* Engaged in strenuous exercise within 5 days of the trial drug administration
* Consumed alcohol within 3 days of the trial drug administration
* Judged as ineligible for the study participation by the investigator for a reason other than above

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2000-07; Primary Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
AUC0-24h (Area under the plasma concentration-time from 0 to 24 hours) | up to 24 hours after drug administration
Cmax (maximum plasma concentration) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 30 days
tmax (time to maximum plasma concentration) | up to 24 hours after drug administration
MRT (Mean residence time) | up to 24 hours after drug administration